CLINICAL TRIAL: NCT03188484
Title: Stepwise High Risk Individuals Screening for Atrial Fibrillation Using Sequential Clinical-electro-biological Register: the AFRICAT Study (Atrial Fibrillation Research In CATalonia)
Brief Title: Atrial Fibrillation Research In CATalonia
Acronym: AFRICAT
Status: Completed | Type: Observational
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Collaborators: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Josep Lluís Clua Espuny, PhD Medicine and Surgery, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Other Study IDs: IDIAP Jordi Gol; 275/C/2015 (Other Grant/Funding Number: FUNDACIO LA MARATO TV3)
Record Dates: First submitted 2017-06-13; First posted 2017-06-15 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Arrhythmia Atrial; Atrial Fibrillation; Hypertension; Diabetes Mellitus
Keywords: Atrial Fibrillation; Electrocardiography; Biological Markers; Risk Assessment
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — A blood sample of 32 cc divided into two serum tubes (8.5 cc), two plasma EDTA tubes (6 cc) and one TempusTM RNA tube (3 cc). Samples will be processed and stored at -20 ºC at the recruiting center until shipment to Neurovascular Research Laboratory, where the sample bank will be set up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The AFRICAT study is a prospective, multicenter, population-based study, which aims to create and apply a sequential screening program for atrial fibrillation (AF) in a high-risk population by integrating clinical, electrocardiographic and biological information. The study will be divided into three different phases of generation, validation and application of a screening program.

In Phase I, from 8,000 individuals aged 65-75 with hypertension and diabetes identified from primary center registries, 100 will be randomly selected . In these patients, the investigators will complete clinical assessment, testing of different pulse-handheld ECG devices (MyDiagnostik, AliveCor and WatchBP) for AF screening, discovery of blood biomarkers for AF (by aptamer technology and RNA expression), and validation of biological candidates from the literature and previous results. All patients will receive Holter monitoring with a wearable device (NuuboTM). In parallel, a predictive risk model for AF will be developed from historical records from the areas in which the study will be carried out.

This Phase I will be followed by a Phase II-validation phase of 400 patients, selected by the predictive model previously mentioned, belonging to the top risk quartile. In these patients, the best biomarkers and devices from phase I will be validated, and patients will be again monitored with the wearable Holter device.

With the results from this validation analysis, a screening program (Phase III) based in the combination of clinical predictors, devices to detect AF (handheld-ECG or pulse wave detectors), blood biomarkers determination and long-term monitoring with wearable Holter. This program will be applied over the whole population targeted by the AFRICAT study, which corresponds to 8,000 patients from 65 to 75 years old, whit hypertension and diabetes mellitus as comorbidities.

DETAILED DESCRIPTION:
The study has been approved by the Ethics Committee of Research Institute IDIAP Jordi Gol (P15/047/2015) and by Hospital Universitari Vall d'Hebron Clinical Research Ethics Committee (PR(AG)133-2015). The study will be conducted in compliance with the Declaration of Helsinki. Registry information was collected from the government-run healthcare provider responsible for all inpatient care in Catalonia. All participants will receive written information and thereafter sign informed consent before inclusion, will be selected among the electronic registers from two different health areas in Catalonia, and will be identified by their 10-digit personal identification number assigned to all citizens in Catalonia.

These patients will be given an appointment in their primary care centre and will receive a comprehensive assessment consisting of:

* Clinical characteristics: demographic factors (age, gender, habits); vascular risk factors (hypertension, diabetes, dyslipidemia), medications, comorbidities (especially those related to AF such as coronary disease, heart failure), vital signs (blood pressure, glycaemia, weight and height).
* Electrocardiographic assessment: three different devices will be tested on each participant (MyDiasnostik, AliveCor and WatchBP). A conventional ECG will be performed to be compared with the results from these devices.
* Blood sample collection: a blood sample of 32 cc divided into two serum tubes (8.5 cc), two plasma EDTA tubes (6 cc) and one TempusTM RNA tube (3 cc). Samples will be processed and stored at -20 ºC at the recruiting centre until shipment to Neurovascular Research Laboratory, where the sample bank will be set up.
* Holter ECG monitoring: a Nuubo Holter will be given to each patient to be carried for four weeks. Electrocardiographic devices will be read blindly. The device records, anonymized and encrypted, will be sent for blinded reading to the Rhythm Disorders Unit from Hospital Virgen del Rocio in Seville.

ELIGIBILITY:
Inclusion Criteria:

All patients aged 65-75 with active diagnoses of hypertension (I10) and diabetes (E10.9 E11.9)

Exclusion Criteria:

* Absence or not accessibility to singular person or its clinical record or/and difficulty to follow the instructions about how managing the devices or/and no acceptation of conditions
* Chronic inflammatory diseases
* Active Cancer
* Dementia
* For Phases II-III: previous diagnosis of AF

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All people included were managed by the Public Health System. Therefore 5,000 participants aged 65-75 with active diagnoses of hypertension (I10) and diabetes (E10.9 E11.9) will be selected from the electronic health record of Primary Care. Given that the registered prevalence of Atrial Fibrillation in this population is was 7.3%, the investigators estimated that around 2.8% will be newly diagnosed with AF at the first study visit. Therefore, the investigators estimate that the number of patients in this population who have undiagnosed AF might be from 140 to 210 patients, taking into account that AF detection should be improved in the study given the long-term monitoring.
Sampling Method: Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation (AF) diagnosis | Study visit/1 month monitoring
  Absence of discrete P waves together with an irregular, arrhythmic pattern of ventricular activation, more than 30 seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Joan Montaner Villalonga, PhD, Study Chair — Neurovascular Research Group
Locations (2):
- Spain (2):
  - SAP Terres de l'Ebre, Tortosa, Tarragona
  - SAP Muntanya, Barcelona

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Abellana R, Gonzalez-Loyola F, Verdu-Rotellar JM, Bustamante A, Pala E, Clua-Espuny JL, Montaner J, Pedrote A, Del Val-Garcia JL, Ribas Segui D, Munoz MA. Predictive model for atrial fibrillation in hypertensive diabetic patients. Eur J Clin Invest. 2021 Dec;51(12):e13633. doi: 10.1111/eci.13633. Epub 2021 Jun 19. PMID 34148231
- [Result] Clua-Espuny JL, Muria-Subirats E, Ballesta-Ors J, Lorman-Carbo B, Clua-Queralt J, Pala E, Lechuga-Duran I, Gentille-Lorente D, Bustamante A, Munoz MA, Montaner J; AFRICAT Research Group. Risk of Atrial Fibrillation, Ischemic Stroke and Cognitive Impairment: Study of a Population Cohort >/=65 Years of Age. Vasc Health Risk Manag. 2020 Oct 28;16:445-454. doi: 10.2147/VHRM.S276477. eCollection 2020. PMID 33149596
- [Result] Garcia-Berrocoso T, Pala E, Consegal M, Piccardi B, Negro A, Gill N, Penalba A, Huerga Encabo H, Fernandez-Cadenas I, Meisel A, Meisel C, Jickling GC, Munoz MA, Clua-Espuny JL, Pedrote A, Pagola J, Juega J, Bustamante A, Montaner J. Cardioembolic Ischemic Stroke Gene Expression Fingerprint in Blood: a Systematic Review and Verification Analysis. Transl Stroke Res. 2020 Jun;11(3):326-336. doi: 10.1007/s12975-019-00730-x. Epub 2019 Sep 2. PMID 31475302
- [Result] Muria-Subirats E, Clua-Espuny JL, Ballesta-Ors J, Lorman-Carbo B, Lechuga-Duran I, Fernandez-Saez J, Pla-Farnos R, On Behalf Members Of Africat Group. Incidence and Risk Assessment for Atrial Fibrillation at 5 Years: Hypertensive Diabetic Retrospective Cohort. Int J Environ Res Public Health. 2020 May 16;17(10):3491. doi: 10.3390/ijerph17103491. PMID 32429492
- [Result] Pala E, Bustamante A, Clua-Espuny JL, Acosta J, Gonzalez-Loyola F, Ballesta-Ors J, Gill N, Caballero A, Pagola J, Pedrote A, Munoz MA, Montaner J. N-Terminal Pro B-Type Natriuretic Peptide's Usefulness for Paroxysmal Atrial Fibrillation Detection Among Populations Carrying Cardiovascular Risk Factors. Front Neurol. 2019 Nov 29;10:1226. doi: 10.3389/fneur.2019.01226. eCollection 2019. PMID 31849809